CLINICAL TRIAL: NCT06539624
Title: A Multicenter, Non-randomized, Open-label, Dose-finding Study to Evaluate the Safety and Preliminary Efficacy of Gene Therapy With EXG110 in Subjects With Fabry Disease
Brief Title: Evaluate the Safety and Preliminary Efficacy of EXG110 in Subjects With Fabry Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Principal Investigator, Mao Jianhua, Vice President of the hospital, The Children's Hospital of Zhejiang University School of Medicine
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EXG110-011
Record Dates: First submitted 2024-07-29; First posted 2024-08-06 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dose escalation-Cohort 1 (Experimental): Genetic : EXG110
  Interventions: Genetic: EXG110 injection
- Dose escalation-Cohort 2 (Experimental): Genetic : EXG110
  Interventions: Genetic: EXG110 injection
- Dose escalation-Cohort 3 (Experimental): Genetic : EXG110
  Interventions: Genetic: EXG110 injection
- Dose escalation-Cohort 4 (Experimental): Genetic : EXG110
  Interventions: Genetic: EXG110 injection

INTERVENTIONS:
Genetic: EXG110 injection — EXG110 is a recombinant adeno-associated virus (rAAV) that not only significantly increases plasma AGA activity, but is also highly expressed in target organs such as the heart and kidneys.EXG110 will be administered in a single dose by intravenous infusion.

SUMMARY:
Objective: To explore the safety and tolerability of different doses of EXG110 with Fabre disease

DETAILED DESCRIPTION:
An open-label, multicenter, single-arm, non-randomized, dose-escalation, and recommended dose-extension clinical design was used to evaluate the safety and efficacy of a single intravenous administration of different doses of EXG110 in patients

ELIGIBILITY:
Inclusion Criteria:

1. At the time of signing the informed consent, age ≥7, male or female
2. Clinical symptoms (at least one Fabry disease related symptom) and genetic diagnosis of Fabry disease,
3. Prior or no prior ERT treatment
4. Have renal or cardiac involvement (adults only)
5. All subjects of reproductive age voluntarily took effective contraception and prohibited sperm donation from entering the screening period until 52 weeks after dosing (main study period)
6. The subjects voluntarily participate and are fully informed, fully understand the research, can comply with the requirements of the research protocol, and are willing to complete the research as planned, and voluntarily provide biological samples for testing according to the requirements of the protocol

Exclusion Criteria:

1. Screening period laboratory test results: a) aspartate aminotransferase or alanine aminotransferase > 1.5× upper limit of normal (ULN);b) Total bilirubin > 1.5× upper limit of normal (ULN);c) Alkaline phosphatase > 2× upper limit of normal (ULN);d) Albumin < lower limit of normal (LLN)
2. There was a clinically significant increase in AFP during the screening period
3. Serum virology test: a) Hepatitis B: Hepatitis B virus surface antigen (HBsAg) positive, and hepatitis B virus-deoxyribonucleic acid (HBV-DNA) higher than the upper limit of normal detection;b) Hepatitis C: if the hepatitis C virus (HCV) antibody is positive, and the hepatitis C virus-ribonucleic acid (HCV-RNA) is higher than the upper limit of normal test value;c) Syphilis: positive for syphilis screening (Tp-Ab) and positive for syphile-specific antibodies;d) HIV: Known human immunodeficiency virus (HIV) positive history or HIV screening positive
4. AVT917 (>1:50), anti-AGA antibody positive(>1:2560)
5. C3 lower than the normal range, C5b-9 higher than the normal range, anti-AVT917 IgM positive
6. Current or have a history of serious cardiovascular disease and surgical history
7. Current underlying liver disease or history of liver disease, as assessed by the investigator, that may affect the safety assessment of the drug
8. Renal disease in adult and the slope of kidney >5 mL/min/1.73m²/year
9. Subjects with poorly controlled diabetes after drug treatment (e.g., HbA1c≥8%);
10. Acute/chronic infection or other chronic disease that the investigator determines will increase the risk of participants participating in the study
11. Patients with a history of malignant tumor or currently suffering from any malignant tumor (except for the following tumor diseases: skin basal cell carcinoma, cervical carcinoma in situ, breast carcinoma in situ, skin squamous cell carcinoma has been controlled after treatment);
12. Have malignancy cancer
13. Patients with active autoimmune diseases (such as rheumatoid arthritis, systemic lupus erythematosus, multiple sclerosis, immune vasculitis, inflammatory bowel disease, etc.);
14. known history of allergy to the components of the investigational products
15. Patients with a history of drug use or drug abuse or alcoholism
16. Use of systemic (intravenous or oral) immunomodulators within the past 6 months or currently
17. Initiation of treatment with blood pressure lowering drugs that affect proteinuria levels (such as angiotensin-converting enzyme inhibitors, angiotensin-receptor blockers, or angiotensin-receptor/enkephalin inhibitors) within 4 weeks prior to screening, or changes in the therapeutic dose of these drugs within 4 weeks prior to screening;
18. Has received, or is currently receiving, a clinical trial of another investigational drug/medical device or treatment (other than vitamins and minerals) within 3 months prior to signing the informed consent (or within 5 half-lives of the investigational drug, whichever is longer)
19. Previous treatment with gene therapy products
20. Those who had received live attenuated vaccine/vaccine within 12 weeks prior to screening or planned to receive it during the study
21. Other clinical conditions that the investigators felt needed to be ruled out

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2027-04-09 (Estimated); Study Completion 2027-04-09 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | 52 weeks following EXG110 administration
  Safety and tolerability of EXG110 following a single IV dose, as assessed by incidence and severity of adverse events, serious adverse events and dose limiting toxicities, including clinically significant changes from baseline to scheduled time points in safety parameters

SECONDARY OUTCOMES:
eGFR change from baseline in mL/min/(1.73m^2); | 52 weeks following EXG110 administration
  eGFR change from baseline in mL/min/(1.73m^2)
NYHA cardiac function grade changed from baseline; | 52 weeks following EXG110 administration
  NYHA cardiac function grade changed from baseline;
Changed from baseline: region and area in mm^2 of skin angiokeratoma The number of Gb3 deposition in skin biopsy under the microscope | 52 weeks following EXG110 administration
  Changed from baseline: region and area in mm^2 of skin angiokeratoma The number of Gb3 deposition in skin biopsy under the microscope
Change from baseline in serum AGA activity | 52 weeks following EXG110 administration
  Change from baseline in serum AGA activity
Change from baseline serum lysoGb3 | 52 weeks following EXG110 administration
  Change from baseline serum lysoGb3

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Mao, PhD, Principal Investigator — Children's Hospital, Zhejiang University School of Medicine
Locations (2):
- China (2):
  - Shanghai Children's Medical Center, Shanghai, Shanghai Municipality
  - Children's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No
All data generated in this study are the property of Hangzhou Jiayin and should be kept strictly confidential together with the information provided by Hangzhou Jiayin.Researchers or any of their staff are not permitted to independently analyze and/or publish these data without the prior written authorization of Hangzhou Jiain.